CLINICAL TRIAL: NCT00795860
Title: Fatty Acid Metabolism and Insulin Sensitivity: the Role of Endurance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: American Diabetes Association (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jeffrey F Horowitz, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ADA - 1-03-JF-10 (completed); ADA grant# 1-03-JF-10 (Other Grant/Funding Number: American Diabetes Association)
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Insulin Resistance and Type 2 Diabetes
Keywords: Insulin sensitivity; fat metabolism; inflammation
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2; Inflammation | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight loss - diet only (Active Comparator)
  Interventions: Behavioral: Weight loss - diet only
- Weight loss plus exercise (Experimental)
  Interventions: Behavioral: Weight loss plus exercise

INTERVENTIONS:
Behavioral: Weight loss - diet only — Subjects adhere to a reduced calorie diet until they lose exactly 12% of their initial body weight. After they achieve this weight loss goal, they are placed on a weight-maintaining diet for 3-4 weeks before follow-up experiments are performed. Subjects meet weekly with a research dietitian throughout their weigh-loss and weight maintenance program.
  Arms: Weight loss - diet only
Behavioral: Weight loss plus exercise — Subjects adhere to a reduced calorie diet and perform 4 session of endurance exercise training per week until they lose exactly 12% of their initial body weight. Exercise training consists of stationary bicycle exercise. the exercise duration and intensity ramp up over the first few weeks of training until subjects exercise 45 min per session at an intensity of 85% of their maximal heart rate. 3 of the 4 exercise session each week are supervised by an Exercise physiologist. After they achieve the 12% weight loss goal, they are placed on a weight-maintaining diet for 3-4 weeks before follow-up experiments are performed. Subjects meet weekly with a research dietitian throughout their weigh-loss and weight maintenance program.
  Arms: Weight loss plus exercise

SUMMARY:
Clearly the effects of diet and exercise are beneficial for obese persons, but the underlying mechanisms for the improvements in metabolic health are not completely clear. Although mounting evidence suggests that alterations in lipid metabolism in persons with abdominal obesity are associated with a several medical complications, including diabetes, little is known about the factors responsible for this effect. The project in this application is designed to examine how the addition of endurance exercise training to a weight-loss program alters whole-body fatty acid availability, uptake, and oxidation as well as the expression of cellular factors that regulate these processes. In addition, we will evaluate whether these alterations are associated with improvements in insulin sensitivity. In the end, these experiments will provide insight into the cellular and whole-body adaptations in fatty acid metabolism in response to weight-loss and exercise training that may lead to enhancement of insulin sensitivity. Identifying relationships between gene expression, whole-body fatty acid metabolism and clinical outcome measurements, such as insulin sensitivity, may lead to improvements in the therapeutic and/or the preventative approach to obesity and its co-morbidities.

DETAILED DESCRIPTION:
Despite robust findings emphasizing the importance of weight-loss and exercise for the prevention and management of insulin resistance and Type 2 diabetes, the mechanisms responsible for the improvements in metabolic health are not completely understood. Mounting evidence suggests that abnormalities in fatty acid metabolism in persons with abdominal obesity are associated with insulin resistance. Alterations in fatty acid mobilization and oxidation may be primary adaptations responsible for the improvements in metabolic health after weight-loss and endurance exercise training. We hypothesize that a disparity between muscle fatty acid uptake and oxidation is regulated by the expression of genes and proteins that participate in intracellular transport, trafficking, and metabolism of fatty acids. We believe that alterations in the expression of these factors in response to weight-loss and endurance exercise training will underlie changes in the non-oxidative disposal of fatty acids, and thereby improve insulin sensitivity. We will determine the effects of weight-loss and exercise training on whole-body fatty acid mobilization and oxidation and the expression of factors that regulate these processes in skeletal muscle. In addition, we will evaluate how these alterations are associated with improvements in insulin sensitivity. These studies will provide insight into how cellular alterations with weight-loss and exercise training and the accompanying changes in whole-body fatty acid metabolism may lead to improvements in metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age = 18-45
* Premenopausal
* Body mass index ≥ 30 kg/m2
* Waist circumference ≥ 100 cm

Exclusion Criteria:

* Evidence of metabolic or cardiovascular disease
* Pregnancy
* Allergies to soybeans or eggs
* Hyperlipidemia (fasting plasma triglyceride concentration > 125 mg/dl)
* Hematocrit < 34%

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2003-06 (Actual); Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | before and after 12% weight loss (3-6 months)

SECONDARY OUTCOMES:
Rate of fatty acid mobilization in plasma | Before and after 12% weight loss (3-6 months)
Abundance and activity of Pro-inflammatory factors in skeletal muscle | Before and after 12% weight loss (3-6 months)
whole body and skeletal muscle oxidative capacity | Before and after 12% weight loss (3-6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Horowitz, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Schenk S, Horowitz JF. Coimmunoprecipitation of FAT/CD36 and CPT I in skeletal muscle increases proportionally with fat oxidation after endurance exercise training. Am J Physiol Endocrinol Metab. 2006 Aug;291(2):E254-60. doi: 10.1152/ajpendo.00051.2006. Epub 2006 May 2. PMID 16670153